CLINICAL TRIAL: NCT06974968
Title: A Phase II Clinical Study Evaluating the Preliminary Efficacy of Human Allogeneic Induced Pluripotent Stem Cell (iPSC)-Derived Motor Neuron Progenitor Cells (XS228 Cell Injection) in Patients With Subacute Spinal Cord Injury
Brief Title: Efficacy of iPSC-Derived Motor Neuron Cells (XS228) in Subacute Spinal Cord Injury: A Phase II Randomized Controlled Trial
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: XellSmart Bio-Pharmaceutical (Suzhou) Co., Ltd. (Industry)
Collaborators: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XS228-Allo-SCI-CN2-P01
Record Dates: First submitted 2025-05-08; First posted 2025-05-16 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-08

CONDITIONS: Spinal Cord Injury; Safety; Efficacy; Clinical Trial; Induced Pluripotent Stem Cells; Human Motor Neuron Progenitor; Transplantation; RCT
Keywords: Spinal Cord Injury; Safety; efficacy; clinical trial; Induced Pluripotent Stem Cells; Human motor neuron progenitor; Transplantation; RCT
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The Phase II study adopts a randomized, double-blind, placebo-controlled design. Investigators and participants remain blinded to treatment allocation. All investigational products and placebos will be identically packaged to maintain blinding for participants, investigators (physicians and coordinators), and monitors. Treatment assignments will remain confidential until database lock and prior to statistical analysis, except in cases of medical emergencies.
  Due to the need for cell-based product preparation based on randomization results, an unblinded team will be established to handle drug preparation and packaging. Unblinded team members will not perform any clinical assessments. Further details are provided in the Drug Management Manual.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- XS228 Interventional Group (Active Comparator): Investigational Product:
  XS228 Cell Injection: Cryopreserved suspension of optimal dose from Phase I. Placebo: Normal saline with identical packaging/labeling. Administration: 4 intrathecal injection via lumbar puncture (Day 1, Day 15, Day 29, Day 43).
  Interventions: Biological: Allogeneic Human Induced Pluripotent Stem Cell (iPSC)-Derived Motor Neuron Progenitor Cells
- Placebo Control Group (Placebo Comparator): Standard rehabilitation protocols
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Allogeneic Human Induced Pluripotent Stem Cell (iPSC)-Derived Motor Neuron Progenitor Cells — Description:
  XS228 Cell Injection is an investigational, allogeneic cell therapy product composed of motor neuron progenitor cells (MNPCs) derived from human induced pluripotent stem cells (iPSCs). This advanced therapy medicinal product (ATMP) is being developed for the treatment of spinal cord injury (SCI) and represents a novel approach in regenerative medicine.
  Arms: XS228 Interventional Group
Other: Placebo — Standard rehabilitation protocols
  Other Names: Standard rehabilitation protocols
  Arms: Placebo Control Group

SUMMARY:
Purpose: This clinical trial is studying an investigational cell therapy called XS228-a lab-made stem cell product designed to help repair damaged nerves in the spinal cord. The goal is to see if XS228 is safe and can improve movement, sensation, and function in people with recent spinal cord injuries.

Study Treatment: XS228 contains specialized nerve-supporting cells derived from human stem cells. These cells are injected into the spinal fluid (intrathecal administration) in a single dose.

Who Can Join? Adults aged 18-65 with a spinal cord injury (thoracic or lumbar level) that occurred 2-12 weeks before enrollment. Participants must have severe but incomplete paralysis (ASIA Impairment Scale Grade A , B or C).

Study Plan:

Phase II (Main Study): About 60 participants will be randomly assigned to receive either XS228 or a placebo (inactive solution) in a 2:1 ratio.

Follow-up: Patients will be monitored for 1 year, with regular check-ups to assess safety, nerve function, and recovery progress.

What Researchers Are Looking For:

Primary Goal: Measure changes in leg and arm function using the ASIA Motor Score at 6 months.

Secondary Goals:

Improvement in ASIA Impairment Scale (AIS) grade (e.g., from "complete" to "incomplete" paralysis).

Recovery of sensation and bladder/bowel control. Safety (monitoring for side effects like infections or immune reactions). Exploratory Tests: MRI scans and biomarker tests in spinal fluid to see if the treatment helps nerve regrowth.

Why This Study Matters: If successful, XS228 could become the first stem cell therapy to promote meaningful recovery in spinal cord injury patients. Currently, no treatments exist to repair nerve damage-this trial aims to change that.

DETAILED DESCRIPTION:
Title: A Randomized, Double-Blind, Placebo-Controlled Phase II Trial to Evaluate the Efficacy and Safety of XS228 Cell Injection in Patients with Subacute Thoracic or Lumbar SCI

Study Type: Interventional (Clinical Trial) Phase: Phase II Allocation: Randomized (2:1, XS228 vs. Placebo) Masking: Double-blind (Participant, Investigator) Primary Purpose: Treatment

Hypothesis:

XS228 (allogeneic iPSC-derived motor neuron progenitor cells) will demonstrate statistically significant improvement in motor function (ASIA Motor Score) compared to placebo at 6 months post-treatment.

The therapy will exhibit an acceptable safety profile with no dose-limiting toxicities (DLTs).

Intervention Details

Investigational Product:

XS228 Cell Injection: Cryopreserved suspension of optimal dose from Phase I. Placebo: Normal saline with identical packaging/labeling. Administration: 4 intrathecal injection via lumbar puncture (Day 1, Day 15, Day 29 and Day 43).

Concomitant Therapies:

Standard rehabilitation protocols (uniform across sites). Prohibited: Other experimental therapies or stem cell treatments during the study.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 65 years (inclusive), regardless of gender.

Etiology: Cervical (C4) to lumbar (L2) spinal cord injury (SCI) caused by traumatic injury or surgery-related factors.

Severity:

Classified as ASIA Impairment Scale (AIS) Grades A, B, or C. MRI-confirmed evidence of spinal cord injury.

Disease Stage:

Primary SCI occurring 14 to 60 days prior to screening (subacute phase).

Contraception:

Participants of childbearing potential (male and female) must agree to use effective non-hormonal contraceptive methods during the trial and for 6 months after trial completion.

Compliance:

Voluntarily participate in the clinical study. Ability to understand and comply with study procedures. Participant or legal guardian can provide written informed consent.

Exclusion Criteria:

* Neurological Inability

Primary spinal cord injury (SCI) during screening with concomitant severe traumatic brain injury precluding neurological function assessment.

Respiratory/Circulatory Instability

High cervical SCI (C1-C3) causing respiratory/circulatory compromise requiring endotracheal intubation or tracheostomy.

Life-Threatening Multiorgan Dysfunction

Concurrent severe injuries to other organ systems with life-threatening dysfunction.

Unstable Thoracoabdominal Injuries

Injuries to lungs, liver, kidneys, spleen, etc., deemed unstable by the investigator.

Prior Spinal Pathology

History of SCI or coexisting spinal disorders (e.g., ankylosing spondylitis, spinal deformities, primary/metastatic spinal tumors, spinal vascular malformations, syringomyelia).

Local Infection/Increased ICP

Active infection at the lumbar puncture site or intracranial hypertension during screening.

Severe Infections

Sepsis, septic shock, or severe pneumonia (per IDSA/ATS 2007 diagnostic criteria).

Confounding Neurological/Psychiatric Conditions

Parkinson's disease, severe dementia, myasthenia gravis, stroke, Guillain-Barré syndrome, diabetic neuropathy, or other conditions interfering with study assessments.

Cardiac Abnormalities (any of the following):

Congestive heart failure (NYHA Class III/IV). Severe uncontrolled arrhythmias (e.g., sick sinus syndrome, third-degree AV block).

Unstable angina or acute myocardial infarction within 3 months prior. Pulmonary Complications

Pulmonary hypertension, pulmonary embolism, or suspected embolism during screening.

Uncontrolled Hypertension/Hypotension

Systolic BP >160 mmHg or diastolic BP >100 mmHg; or systolic BP <90 mmHg or diastolic BP <60 mmHg.

Active Autoimmune Diseases

Requiring immunosuppressants (e.g., uncontrolled hyperthyroidism, systemic lupus erythematosus).

Immunosuppressant Non-Compliance

Unwillingness or inability to use immunosuppressants per protocol.

Laboratory Abnormalities (any of the following):

ALT/AST >2×ULN or total bilirubin >2×ULN. eGFR <60 mL/min/1.73m² (CKD-EPI 2021 formula). APTT/PT >2.5×ULN (without anticoagulants). Platelets <100×10⁹/L or hemoglobin <90 g/L. Allergy

History of severe allergies or hypersensitivity to trial drug/excipients (human albumin, lactated Ringer's solution).

Infectious Diseases

HBsAg+ with HBV DNA >1000 IU/mL; HCV-Ab+; HIV-Ab+; or TP-Ab+. Lumbar Puncture Refusal

Unwillingness to undergo intrathecal administration procedures. Pregnancy/Lactation

Females who are pregnant or breastfeeding. Malignancy

Active malignancy or anticancer therapy within 5 years prior. Recent Clinical Trial Participation

Enrollment in another drug trial within 3 months prior. Investigator Discretion

Any condition deemed unsuitable for participation by the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2028-05-25 (Estimated); Primary Completion 2031-05-25 (Estimated); Study Completion 2031-05-26 (Estimated)

PRIMARY OUTCOMES:
Improvement in ASIA Impairment Scale (AIS) grade | Improvement in ASIA Impairment Scale (AIS) grade from baseline at Day 29, Day 90, Day 180, Day 270, and Day 360 after the first dose administration.

SECONDARY OUTCOMES:
Changes in American Spinal Injury Association (ASIA) Motor Score | From baseline at Day 29, Day 90, Day 180, Day 270, and Day 360 after the first dose administration.
  Changes in motor scores assessed by the ASIA score scale (total score range from 0 to 100, higher values represent a better outcome)
Changes in American Spinal Injury Association (ASIA) Sensory Score | From baseline at Day 29, Day 90, Day 180, Day 270, and Day 360 after the first dose administration.
  Changes in sensory scores assessed by the ASIA score scale (total score range from 0 to 224, higher values represent a better outcome)
Changes in Spinal Cord Independence Measure-III (SCIM-III) | From baseline at Day 29, Day 90, Day 180, Day 270, and Day 360 after the first dose administration.
  SCIM-III(range: 0-100, with lower score indicating greater disability)
Safety and Tolerability | From baseline at Day 29, Day 90, Day 180, Day 270, and Day 360 after the first dose administration.
  Description: Systematic evaluation of:
  Adverse events (AEs) up to 360 days post-infusion Immunogenicity (anti-HLA antibodies, T-cell responses)
  Assessment Methods:
  CTCAE v5.0 grading Neurological monitoring (ISNCSCI exams) CSF analysis for inflammation markers

CONTACTS AND LOCATIONS:
Overall Officials: Limin Rong, prof and M.D, Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
At this stage, the sponsor has not yet finalized a decision regarding the sharing of individual participant data (IPD). The potential risks and benefits of data sharing, including patient privacy, regulatory requirements, and intellectual property considerations, are still under evaluation. A final determination will be made following further internal review and alignment with applicable data protection laws, institutional policies, and ethical guidelines. If IPD sharing is approved in the future, details regarding data accessibility, anonymization methods, and request procedures will be specified in an updated plan.